CLINICAL TRIAL: NCT04073251
Title: Randomized, Controlled, Double Blind Clinical Study on the Assessment of Efficacy, Safety and Palatability of "KalobaTuss® Children", a Syrup for the Treatment of Cough in Pediatric Age (3-6 Years).
Brief Title: Efficacy, Safety and Palatability of the Syrup "KalobaTuss® Children" for the Treatment of Cough in Children
Acronym: KALOCOUGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Principal Investigator, Gioacchino Calapai, FULL PROFESSOR OF PHARMACOLOGY AND TOXICOLOGY, Azienda Ospedaliera Universitaria Policlinico "G. Martino"
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KTC
Record Dates: First submitted 2019-08-19; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Cough
Keywords: Persistent cough; Children
MeSH Terms: conditions — Cough; Chronic Cough

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind controlled clinical study .
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KalobaTuss children (Experimental): KalobaTuss children syrup 5 ml for 4 times a day supplied for 8 consecutive days.
  Interventions: Dietary Supplement: KalobaTuss children
- Placebo (Placebo Comparator): Placebo syrup 5 ml for 4 times a day supplied for 8 consecutive days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: KalobaTuss children — Syrup, dosage: 5 ml for 4 times a day for 8 days.
  Arms: KalobaTuss children
Dietary Supplement: Placebo — Syrup, dosage: 5 ml for 4 times a day for 8 days.
  Arms: Placebo

SUMMARY:
Cough of children is one of the most frequent events for which parents ask for a medical consult and it is a true challenge for pediatrics during daily practice.

In the majority of cases, it is self-limiting, but its persistence could become exasperating and it could reduce quality of life and social activities.

Even if inappropriate prescription of antitussive pharmacological treatment in children has been reduced, pediatrics prescribing attitudes do not still always are reflecting accurate treatment of cough.

Furthermore, pediatric approach is always compromised by parental exaggerate perception of symptoms and usual consequent requirement of pharmacological prescription of antibiotics, that they consider the appropriate and effective therapeutic option for cough.

The World Health Organization identifies honey as a potential demulcent treatment for cough.

On the light of the above considerations and since available pediatric treatments for acute cough are limited by lack of demonstrated efficacy, a pediatric cough syrup product containing Acacia honey as well as specific fractions of resins, polysaccharides, saponins, flavonoids and sugars derived from Malva sylvestris extract, Inula helenium, Plantago major extract, Helichrysum stoechas (KalobaTuss) was developed to be clinically tested on persisting cough of children. Investigators evaluated through a randomized, double blind controlled clinical study the effects of KalobaTuss on persistent cough in children aging 3-6 years. The effects of Kalobatuss were compared with effects of placebo on nocturnal and daytime persistent cough for eight days. Objective of the study was to evaluate the clinical efficacy of KalobaTuss by using as primary endpoint the assessment of changes in day- and night-time cough score.

DETAILED DESCRIPTION:
Cough of children is one of the most frequent events for which parents ask for a medical consult and it is a true challenge for pediatrics during daily practice. Cough is perhaps the most troubling symptom for children suffering from upper respiratory tract infections (URIs) and their parents. Often It results in discomfort to the child and loss of sleep for both children and parents.

In the majority of cases, persistent cough is self-limiting, but its persistence could become exasperating and it could reduce quality of life and social activities.

The influence of persistent cough of children on family's life can create growing discomfort. Indeed, children with acute cough may experience transient disability which leads to lose parents' work and school days so increasing overall cost for its management. Generally, parents' concerns increase when children's cough lasts for more than a week. Consequently, often occurs that parents seek for a medical consult with requirement of drug treatment, even if the most of antitussive drugs lack of proved evidence of effectiveness and safety.

Even if inappropriate prescription of antitussive pharmacological treatment in children has been reduced, pediatrics prescribing attitudes do not still always are reflecting accurate treatment of cough.

Furthermore, pediatric approach is always compromised by parental exaggerate perception of symptoms and usual consequent requirement of pharmacological prescription of antibiotics, that they consider the appropriate and effective therapeutic option for cough. Epidemiological data indicate that cough in children is much more feared than in adults and a substantial proportion of individuals think of cough as "a disease". Also a recent Italian survey confirms this view by suggesting that some pediatricians' therapeutic attitudes should be substantially improved in order to achieve better management of cough in children and to minimize the burden of cough. Moreover, it often happens that attempting to treat cough, children are administered with over-the-counter products having little or no scientific evidence of proven efficacy.

The World Health Organization identifies honey as a potential demulcent treatment for cough. Administration of honey before bedtime has been reported by parents as being preferable to dextromethorphan, diphenhydramine or placebo for symptomatic relief of their child's nocturnal cough and sleeping difficulty due to URIs. A separate clinical entity is cough when is without an organic cause. Such a persistent involuntary cough without a cause is considered to be a functional disorder.

On the light of the above considerations and since available pediatric treatments for acute cough are limited by lack of demonstrated efficacy, a pediatric cough syrup product containing Acacia honey as well as specific fractions of resins, polysaccharides, saponins, flavonoids and sugars derived from Malva sylvestris extract, Inula helenium, Plantago major extract, Helichrysum stoechas (KalobaTuss) to be clinically tested on persisting cough of children, has been developed. Researchers investigated through a randomized, double blind controlled clinical study the effects of KalobaTuss or placebo on persistent cough in children aging 3-6 years. Aim of this trial is to compare the effects of Kalobatuss with effects of placebo on nocturnal and daytime persistent cough for eight days.

Methods This randomized, double-blind controlled clinical study was carried out in the pediatric consulting rooms of the Azienda Ospedaliera Provinciale of Messina together with the Azienda ospedaliera Universitaria Policlinico "G. Martino of Messina, Italy. Children recruited for the study were divided in two groups: children belonging to the active group received the syrup KalobaTuss and the second group received a placebo as syrup formulation. Randomization was performed according to a table generated by Excel program. The double-blinding was released and the treatment groups to be revealed only after the analysis of the study results. Children aged between 3 and 6 years, with persistent cough for at least three consecutive days, which led parents to the need for medical consultation, participated in the study. Children with history of obstructive pulmonary diseases, cystic fibrosis, neuropathies, heart disease, diabetes and immunodeficiencies were excluded. Children suitable according to the inclusion criteria were randomly assigned to one of the treatment groups (KalobaTuss or placebo). Parents or tutors according children participation signed the informed consent form. The two treatment regimens were administered 4 doses a day, 5 ml each, for 8 days. The appearance, consistency, organoleptic characteristics and viscosity of KalobaTuss and placebo were similar.

The study was approved by the Ethic Committee of Azienda Ospedaliera Universitaria Policlinico "G. Martino" with protocol number 95/18 on 17 December 2018. The trial was conducted according to the ethical principles of the Seoul revision (2008) of the Helsinki Declaration and Good Clinical Practice.

Objective of the study was to evaluate the clinical efficacy of KalobaTuss by using as primary endpoint the evaluation and analysis of changes in day- and night-time cough score assessed through a questionnaire filled by parents. Cough was clinically diagnosed and evaluated by the pediatrician during the first visit and successively monitored by parents by filling a daily diary. At the end of the administration period pediatrician visited again children and collected the daily diary for each child.

The sample size was obtained assuming a mean cough score of 3 points in both groups at baseline, and a mean change in cough score of 2 and 1 points respectively for the arm treated with the study product and the placebo arm.

110 children with persistent cough were enrolled, 106 (96.36%) completed the treatment. 54 children received the KalobaTuss syrup and another 52 children received the placebo syrup. Four children, two from each group, left the study before the end of treatment.

The median age of children completing the study was 53.02 ± 12.02 months (range, 38-70 months; median age 4.3 months), with no significant difference in age between the two treatment arms (p= 0.8181).

54 children (50.8 %) were boys, of which 28 (51.85%) in the KalobaTuss syrup arm and 26 (48.15%) in the placebo arm. The mean duration of coughing before enrollment was 3.53 ± 0.57 (SD) for the KalobaTuss syrup and 3.52 ± 0.58 (SD) for the placebo arm, with no significant difference between the two arms (P= 0.93624). None of the children monitored for the study needed to receive antibiotics or any other pharmacological therapy during the days of treatment and for the follow-up period of one week after the end of the study.

Adverse events (AEs) were monitored during all the study period. An AE was defined as an inconvenient medical event occurring during the study period whether or not it was linked to the study procedure or the study product. A severe AE (SAE) was defined as a medical event resulting in death, a life-threatening situation, requiring inpatient admission or prolongation of hospitalization, and/or resulting in severe or persistent subject disability or incapacity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged between 3 and 6 years, with persistent cough for at least three consecutive days.

Exclusion Criteria:

* Children with history of obstructive pulmonary diseases, cystic fibrosis, neuropathies, heart disease, diabetes and immunodeficiencies were excluded.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Assessment of efficacy of treatment of cough persistent | 8 weeks
  Primary endpoint is the assessment of changes in day- and night-time cough score. Cough was diagnosed and evaluated by the pediatrician during the first visit and monitored by parents by filling a daily diary. At the end of the administration period pediatrician visited again children and collected the daily diary for each child.

CONTACTS AND LOCATIONS:
Overall Officials: Gioacchino Calapai, MD, Principal Investigator — Azienda Ospedaliera Universitaria "G Martino", Messina, Italy.
Locations (1):
- Gioacchino Calapai, Messina, Me, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Blasio F, Dicpinigaitis PV, Rubin BK, De Danieli G, Lanata L, Zanasi A. An observational study on cough in children: epidemiology, impact on quality of sleep and treatment outcome. Cough. 2012 Jan 23;8(1):1. doi: 10.1186/1745-9974-8-1. PMID 22269875
- [Background] Zanasi A, Morcaldi L, Cazzato S, Mazzolini M, Lecchi M, Morselli-Labate AM, Mastroroberto M, Dal Negro RW. Survey on attitudes of Italian pediatricians toward cough. Clinicoecon Outcomes Res. 2017 Mar 16;9:189-199. doi: 10.2147/CEOR.S129696. eCollection 2017. PMID 28352199
- [Background] French CT, Irwin RS, Fletcher KE, Adams TM. Evaluation of a cough-specific quality-of-life questionnaire. Chest. 2002 Apr;121(4):1123-31. doi: 10.1378/chest.121.4.1123. PMID 11948042
- [Background] Dal Negro RW, Mazzolini M, Turco P, Zanasi A. Cough: impact, beliefs, and expectations from a national survey. Multidiscip Respir Med. 2016 Sep 27;11:34. doi: 10.1186/s40248-016-0072-1. eCollection 2016. PMID 27708777
- [Background] Rousounidis A, Papaevangelou V, Hadjipanayis A, Panagakou S, Theodoridou M, Syrogiannopoulos G, Hadjichristodoulou C. Descriptive study on parents' knowledge, attitudes and practices on antibiotic use and misuse in children with upper respiratory tract infections in Cyprus. Int J Environ Res Public Health. 2011 Aug;8(8):3246-62. doi: 10.3390/ijerph8083246. Epub 2011 Aug 5. PMID 21909304
- [Background] Smith SM, Schroeder K, Fahey T. Over-the-counter (OTC) medications for acute cough in children and adults in community settings. Cochrane Database Syst Rev. 2014 Nov 24;2014(11):CD001831. doi: 10.1002/14651858.CD001831.pub5. PMID 25420096
- [Background] Paul IM, Beiler J, McMonagle A, Shaffer ML, Duda L, Berlin CM Jr. Effect of honey, dextromethorphan, and no treatment on nocturnal cough and sleep quality for coughing children and their parents. Arch Pediatr Adolesc Med. 2007 Dec;161(12):1140-6. doi: 10.1001/archpedi.161.12.1140. PMID 18056558
- [Background] Cohen HA, Rozen J, Kristal H, Laks Y, Berkovitch M, Uziel Y, Kozer E, Pomeranz A, Efrat H. Effect of honey on nocturnal cough and sleep quality: a double-blind, randomized, placebo-controlled study. Pediatrics. 2012 Sep;130(3):465-71. doi: 10.1542/peds.2011-3075. Epub 2012 Aug 6. PMID 22869830
- [Background] Chung KF. Assessment and measurement of cough: the value of new tools. Pulm Pharmacol Ther. 2002;15(3):267-72. doi: 10.1006/pupt.2002.0360. PMID 12099776
- [Background] Weinberger M, Lockshin B. When is cough functional, and how should it be treated? Breathe (Sheff). 2017 Mar;13(1):22-30. doi: 10.1183/20734735.015216. PMID 28289448
- [Derived] Carnevali I, La Paglia R, Pauletto L, Raso F, Testa M, Mannucci C, Sorbara EE, Calapai G. Efficacy and safety of the syrup "KalobaTUSS(R)" as a treatment for cough in children: a randomized, double blind, placebo-controlled clinical trial. BMC Pediatr. 2021 Jan 11;21(1):29. doi: 10.1186/s12887-020-02490-2. PMID 33430841